CLINICAL TRIAL: NCT07186920
Title: Lung Ultrasound Assessment of Postoperative Atelectasis After Mechanical Ventilation With Minimum Driving Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University General Hospital of Patras (Other)
Responsible Party: Principal Investigator, Antonios Kostouros, Anesthesiology Resident, Antonios Kostouros, University General Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22623 / 4.8.2025
Record Dates: First submitted 2025-08-20; First posted 2025-09-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Atelectasis; Postoperative Pulmonary Atelectasis; Postoperative Pulmonary Complications (PPCs); Lung Ultrasonography Score; Lung Ultrasound
Keywords: Postoperative Atelectasis; Postoperative Pulmonary Atelectasis; Postoperative pulmonary complications (PPCs); Lung ultrasonography score; Lung ultrasound; Atelectasis; Pulmonary atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung Protective Ventilation (Other): CONVENTIONAL LUNG PROTECTIVE VENTILATION
  This group is mechanically ventilated with Invasive Mechanical Ventilation with PEEP 8 cm H20 Tidal Volume (VT) 8 ml/kg Ideal Body Weight (IBW) Respiratory Rate (RR) --> PaCO2 = 35-45 mmHg Inspired Oxygen Fraction (FiO2) 0.4 - 0.5 --> Pulse Saturation Oxygen (SpO2) > 93% Recruitment Maneuver (as described) every hour
  Interventions: Procedure: Lung Protective Ventilation
- Minimum Driving Pressure (Active Comparator): This group is mechanically ventilated with Invasive Mechanical Ventilation with PEEP; Initially 8 cm H20, titrated at level with Minimum Driving Pressure after first recruitment - titration maneuver followed by new recruitment maneuver VT 8 ml/kg IBW RR --> PaCO2 = 35-45 mmHg FiO2 0.4 - 0.5 --> SpO2 > 93% Recruitment Maneuver (as described) every hour
  Interventions: Procedure: PEEP titration for Minimum Driving Pressure

INTERVENTIONS:
Procedure: PEEP titration for Minimum Driving Pressure — This group is mechanically ventilated with Invasive Mechanical Ventilation with Volume Control Ventilation mode with PEEP Initially 8 cm H2O. Afterwards, the lungs are recruited with the aforementioned maneuver. During subsequent derecruitment, PEEP is decreased by 2 cm H20 and compliance is noted in each stage. The goal is to find PEEP with maximum compliance (Cmax). A new recruitment maneuver follows and during derecruitment PEEP is set at the optimum value that was previously defined.
  VT 8 ml/kg IBW RR --> PaCO2 = 35-45 mmHg FiO2 0.4 - 0.5 --> SpO2 > 93% Recruitment Maneuver (as described) every hour
  Other Names: Maximum compliance mechanical ventilation; Cmax Mechanical Ventilation
  Arms: Minimum Driving Pressure
Procedure: Lung Protective Ventilation — This group is mechanically ventilated with Invasive Mechanical Ventilation with Volume Control Ventilation mode with PEEP 8 cm H2O. VT 8 ml/kg IBW RR --> PaCO2 = 35-45 mmHg FiO2 0.4 - 0.5 --> SpO2 > 93% Recruitment Maneuvers (as described) every hour
  Arms: Lung Protective Ventilation

SUMMARY:
Brief summary The goal of this clinical trial is to compare two different types of perioperative mechanical ventilation (MV), specifically Protective Mechanical Ventilation (PMV) and MV with the lowest possible Driving Pressure (ΔP), in relation to the appearance of postoperative lung closing, eg atelectasis, in adult patients who are operated. Atelectasis will be evaluated via lung ultrasound.

The main questions it aims to answer are:

* Is MV with lower ΔP better than conventional PMV in keeping lungs more open perioperatively and immediately postoperatively?
* Does MV with lower ΔP decrease hospital stay, Intensive Care Unit (ICU) need and mortality?

Researchers will use lung ultrasound to compare MV with the lowest possible Driving Pressure (ΔP) to Protective Mechanical Ventilation (PMV) to see if any of this is more protective than the other concerning lung atelectasis.

All participants will receive perioperative MV.

Half of them will receive conventional Protective Mechanical Ventilation (PMV). This will include well known generally protective settings for mechanical ventilation of patients, concerning volumes, pressures, respiratory rate, inspiratory gases and ventilation maneuvers.

The rest of participants will be ventilated with the lowest possible Driving Pressure (ΔP). This will be similar to PMV in the chosen volumes, respiratory rate, inspiratory gases and ventilation maneuvers. However, the pressure inside lung at the end of expiration, eg Positive End Expiratory Pressure (PEEP), will be not be preset for every patient. Initially, we will perform a maneuver that will quantify each individual's lung characteristics and mechanics. According to this, we will find the exact PEEP that seems to suit each patients lungs most, and use this perioperatively, trying to provide lungs the best conditions every time.

After the completion of the operation, all the patients will be screened for atelectasis, via lung ultrasound, using a well established protocol for the quantification of atelectasis. The results will be statistically analyzed trying to find if any of the forementioned strategies of mechanical ventilation surpasses the other concerning atelectasis appearance.

Furthermore efficiency of lung oxygen absorption, hospital stay, ICU need and mortality will be noted.

ELIGIBILITY:
Inclusion Criteria:

* >17 years old
* Surgery with general anesthesia & invasive mechanical ventilation
* ASA score I-III

Exclusion Criteria:

* <18 years old
* Preoperative ARISCAT score estimation <26
* Women during pregnancy or just given birth
* Other type of anesthesia (Not general)
* Contraindication of administration of neuromuscular blockade agents.
* Contraindication of cease of spontaneous ventilation.
* Mechanical ventilation without endotracheal intubation.
* Severe heart failure / History of ischemic heart disease.
* Moderate or severe chronic obstructive lung disease or interstitial lung disease.
* History of operation in heart, lung or diaphragm.
* Presence of new active pathology in respiratory system at the beginning of surgery (infection / trauma / anatomic disorder).
* Severe intraoperative respiratory complication (laryngospasm / bronchospasm / anaphylaxis).
* Immediate postoperative need for continuation of IMV.
* Patient denial of participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-10-06 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Lung Ultrasound Score (LUS) | Within 20 minutes in PACU.
  12 Position Lung Ultrasound will be performed in Post Anesthesia Care Unit (PACU) within 20 minutes postoperatively. In each position the potential scores will be 0,1,2 and 3.
  0 --> 0-2 B-lines
  1. --> >2 B-lines or presence of small sublpleural consolidations with normal pleural line.
  2. --> Multiple coalescent B-lines or multiple small sublpleural consolidations with thickened or irregular pleural line.
  3. --> Total air loss or subpleural consolidation with diameter bigger than 1x2cm. The total sum of ultrasound scores of each position is marked as LUS.

SECONDARY OUTCOMES:
Rate of Postoperative Respiratory Failure | Within 30 minutes in PACU
  Postoperative Respiratory Failure based on Arterial Blood Gases in PACU (type I and/or II) Type I --> Arterial Oxygen Partial Pressure / Arterial Oxygen Saturation (P/F) ratio <300 Type II --> PaCO2 > 45mmHg
Rate of NIMV need | Period of stay in Post Anesthesia Care Unit (PACU). From time of postoperative transfer to PACU until time of discharge from PACU and return to general clinic, an average of 1 hour.
  Potential need for NIMV in PACU due to Respiratory Failure.
  CPAP / BIPAP / High-Flow Nasal Canula
Hospital Stay | From day of operation until the end of patient stay inside hospital, because of return to home or due to death.
  Total hospital stay days from day of operation until hospital discharge.
ICU need. | From day of operation until the end of patient stay inside hospital, because of return to home or due to death.
  Potential Need for ICU admission.
ICU stay | From day of operation until the end of patient stay inside hospital, because of return to home or due to death.
  In case of ICU need, total days of ICU stay.
28 Day mortality | From day of operation until up to 28 days.
  Incidence of death in 28 days in each group.
Mechanical Power (MP) | From the moment of beginning of operation until the moment of the end of operation and mechanical ventilation
  o To calculate MP, the following must be recorded: RR, Peak Airway Pressure (Ppeak), Plateau Pressure (Pplat), and PEEP. The simplified equation will be used; MP = 0.098 × RR × [Ppeak - (Plat-PEEP)/2]
Volume-normalized Mechanical Power (MPcrs) | From the moment of beginning of operation until the moment of the end of operation and mechanical ventilation
  MPcrs = MP/Respiratory System Compliance (Crs)
Elastic Power (EP) | From the moment of beginning of operation until the moment of the end of operation and mechanical ventilation
  To calculate EP, the following must be recorded: RR, VT, Pplat, and PEEP. The following equation will be used:
  EP = 0.098 × RR × VT × [(Plat+PEEP)/2]
Volume-normalized Elastic Power (EPcrs) | From the moment of beginning of operation until the moment of the end of operation and mechanical ventilation
  EPcrs = EP/Crs

CONTACTS AND LOCATIONS:
Overall Officials: Diamanto Aretha, A. Professor, Study Chair — University of Patras; Nektaria Xirouchaki, Consultant, Study Director — University of Crete; Eumorfia Kondili, Professor, Study Director — University of Crete; Antonios Kostouros, Resident, Principal Investigator — University of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: Yes